CLINICAL TRIAL: NCT00308529
Title: Phase II Study of Irinotecan, Carboplatin, Bevacizumab, and Radiation Therapy in the Treatment of Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Irinotecan, Carboplatin, Bevacizumab, and Radiation Therapy in the Treatment of Limited Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 110; AVF3526s
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-01

CONDITIONS: Carcinoma, Small Cell Lung; Lung Cancer
Keywords: Carcinoma Small Cell Lung; Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Irinotecan; Carboplatin; Bevacizumab; Radiotherapy

INTERVENTIONS:
Drug: irinotecan
Drug: carboplatin
Drug: bevacizumab
Procedure: Radiation Therapy

SUMMARY:
This proposed phase II trial will investigate the combination of irinotecan, carboplatin and bevacizumab along with radiation in the treatment of patients with limited-stage SCLC. This study differs from our "maintenance" bevacizumab trial in that bevacizumab will begin with the initial chemotherapy treatment. Irinotecan/platinum regimens are emerging as standard treatments for patients with extensive-stage disease. Adding a novel minimally toxic agent to this regimen up front may further enhance this doublet's efficacy without contributing to toxicity. This trial will be one of the first clinical trials to evaluate a combination of targeted therapy and chemotherapy in the up front treatment of a common solid tumor.

DETAILED DESCRIPTION:
Eligible patients will receive 4 courses of irinotecan, carboplatin, and bevacizumab. Radiation therapy will begin concurrently with the third course of systemic treatment. The intervals between chemotherapy courses will be 28 days.Patients will be completely restaged approximately 2 weeks after completion of chemotherapy prior to beginning treatment with maintenance bevacizumab. Those with progressive tumor or serious toxicity will come off study. Those with stable disease or objective tumor responses will continue treatment with restaging every 12 weeks for a minimum of 6 cycles (6 months).

* Induction chemotherapy regimen Irinotecan: 60mg/m2 IV on days 1, 8, and 15 Carboplatin: AUC=4 day 1 only Bevacizumab 10 mg/kg IV days 1, 15 Cycles are repeated every 28 days for four courses
* Radiation therapy 1.8 Gy, single daily fractions, concurrently with the third course of chemotherapy e to a total dose of 61.2 Gy (34 fractions). Patients obtaining complete remission or near complete remission will also receive prophylactic whole brain radiotherapy, given within one month after all therapy is completed (total dose 24Gy in 2Gy daily fractions).
* Maintenance Bevacizumab Bevacizumab alone at a dose of 10 mg/kg IV days 1 and 15 each cycle, for a maximum of 6 additional cycles (6 months) with restaging every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed small cell lung cancer.
* Limited stage disease (
* ECOG performance status 0 or 1.
* No previous treatment with chemotherapy, radiation therapy, or biologic agents.
* Measurable disease
* Adequate bone marrow, liver, kidney function
* Patients must be able to understand the nature of this study and give written consent.

Exclusion Criteria:

* Age < 18 years
* History of a prior malignancy within three years with the exception of skin cancer (excluding melanoma), cervical carcinoma in situ, in situ breast carcinoma, or early stage prostate cancer.
* Women who are pregnant or lactating are ineligible. Men and women of childbearing potential are required to use adequate contraception during this study.
* History or physical exam evidence of CNS disease (eg seizures not controlled with standard medical therapy, history of stroke)
* Active infection requiring parenteral antibiotics
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or fine needle aspiration within 7 days of beginning bevacizumab or anticipation of need for major surgical procedure during the course of the study.
* Full-dose oral or parenteral anticoagulation must be on a stable dosing schedule prior to enrollment.
* Proteinuria
* Serious nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Prior hemoptysis.
* History of acute myocardial infarction or stroke within 6 months
* Uncontrolled hypertension (> 150/100), unstable angina, New York Heart Association grade II or greater CHF, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease.
* Received other investigational drugs within 28 days
* PEG, G-tubes, or other percutaneous drains/tubes
* History of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or place the subject at high risk for treatment complications
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2006-03; Primary Completion 2007-04 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
progression-free survival

SECONDARY OUTCOMES:
toxicity
overall response rate
duration of response
overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (4):
- United States (4):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Hainsworth JD, Yardley DA, Raefsky E, Patton J, Peacock N, Farley C, Burris HA 3rd, Greco FA. Tracheoesophageal fistula formation in patients with lung cancer treated with chemoradiation and bevacizumab. J Clin Oncol. 2010 Jan 1;28(1):43-8. doi: 10.1200/JCO.2009.24.7353. Epub 2009 Nov 9. PMID 19901100